CLINICAL TRIAL: NCT04825392
Title: A Phase Ib Study of Tolerance and Safety of a Recombinant Anti-PD-1 Monoclonal Antibody HX008 in Patients With Advanced Solid Tumors
Brief Title: A Phase Ib Study of HX008 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou Hanzhong biomedical co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX008-Ib-01
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HX008 (Experimental)
  Interventions: Drug: HX008

INTERVENTIONS:
Drug: HX008 — Patients will receive HX008 3mg/kg by intravenous (IV) infusion on Day 1, every 3 weeks (Q3W), till progressed disease or withdrawal.

SUMMARY:
HX008 is a humanized monoclonal antibody targeting PD-1 on the T cell surface, restores T cell activity, thus enhancing immune response, and has the potential to treat various types of tumors. In this study, the tolerance and safety of HX008 in patients with advanced solid tumors will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent voluntarily. Understand this protocol and be willing and able to adhere to the study visit schedule;
* Male and Female aged ≥18 are eligible;
* Patients with locally advanced or metastatic solid tumors confirmed by histology or cytology, progressed after the failure of standard treatment, or could not accept/have no standard treatment;
* The patients with ECOG score of 0 or 1;
* The expected survival time is at least 3 months;
* Subjects should have measurable lesions (at least one extracranial lesion) According to RECIST v1.1;
* If the subjects received anti-tumor treatment, they need to meet the following conditions:

The interval between whole-body radiotherapy and the first administration in this study was more than 3 weeks, and the interval between local radiotherapy or radiotherapy for bone metastasis and the first administration was more than 2 weeks. No radiopharmaceuticals were taken within 8 weeks before the first administration. The interval between previous chemotherapy or targeted therapy and the first administration of this trial was ≥ 4 weeks or the interval was ≥ 5 half-lives (whichever occurs first); The interval between immunotherapy or biotherapy (tumor vaccine, cytokine, or growth factor controlling cancer) and the first administration of this study was more than 6 weeks;

* Has sufficient organ and bone marrow function to meet the following laboratory examination standards:

  1. Blood routine: absolute neutrophil count (ANC)≥1.5×10^9/L; white blood cell count (WBC)≥3×10^9/L; platelet count (PLT)≥100×10^9/ L; hemoglobin (HGB)≥90 g/L;
  2. Renal function: Serum creatinine (Scr) ≤1.5×ULN;
  3. Liver function: TBIL≤1.5×ULN; Patients without liver metastases require alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5× ULN. Patients with liver metastases require ALT and AST≤5×ULN;
  4. The coagulation function is adequate, which is defined as the international normalized ratio (INR) ≤ 2×ULN; or activated partial thromboplastin time (APTT)≤ 1.5×ULN;
* Reproductive men and women of childbearing age are willing to take effective contraceptive measures from signing the informed consent form to 3 months after the last administration of the trial drug.

Exclusion Criteria:

* Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as carcinoma in situ of the cervix or basal cell skin cancer;
* With adverse reactions of previous treatment that have not recovered to CTCAE V5.0 grade ≤ 1, except for the residual hair loss effect;
* Prior treatment with anti-PD-1/PD-L1/CTLA-4 antibody;
* With active or history of autoimmune diseases that may recur (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulitis, etc.), or patients with high risk (e.g., organ transplantation requiring immunosuppressive therapy). While those with the following diseases were allowed to be enrolled: a) Stable patients with type I diabetes after a fixed dose of insulin; b) Autoimmune hypothyroidism requiring hormone replacement therapy only; c) Skin diseases requiring no systemic treatment (e.g. eczema, skin rash covering less than 10% of the body surface, psoriasis without ophthalmic symptoms, etc.);
* Expecting to receive major surgery during the study period including 4 weeks prior to the first dose of the study drug;
* Need to receive systemic corticosteroids (dose equivalent to > 10 mg prednisone/day) or other immunosuppressive drugs within 14 days before enrollment or during the study period. Those under the following conditions are eligible: a) Locally external use or inhaled corticosteroids; b) short-term (≤ 7 days) use of glucocorticoids for the prevention or treatment of nonautoimmune allergic diseases;
* Suffered from idiopathic lung disease, interstitial lung disease, pulmonary fibrosis, acute lung disease, etc., except for local interstitial pneumonia induced by radiotherapy;
* Has uncontrolled systemic diseases, for instance, cardiovascular and cerebrovascular disease, diabetes, tuberculosis;
* History of human immunodeficiency virus infection, acquired or congenital immunodeficiency disease, organ transplantation, or stem cell transplantation;
* Patients with symptomatic central nervous system metastasis (patients with asymptomatic central nervous system metastasis or asymptomatic brain metastasis after treatment, without disease progression by CT / MRI examination, and with a time interval of more than 4 weeks from the last radiotherapy are eligible.);
* Patients with active tuberculosis;
* Patients with chronic hepatitis B or active hepatitis C. Except for Hepatitis B virus carriers or those with stable hepatitis B after drug treatment with DNA titer no higher than 500 IU/ml or copy number < 1000 copies/ml, and cured hepatitis C patients (HCV RNA test negative);
* Has severe infection within 4 weeks or active infection requiring IV infusion of antibiotics within 2 weeks prior to the first dose of the study drug;
* Known to be allergic to macromolecular protein agents or monoclonal antibodies. Known to has a history of severe allergies to any of the components in the study drug (CTCAE v5.0 ≥ grade 3);
* Has participated in other clinical trials within 4 weeks prior to the first dose of the study drug;
* Alcohol dependence or drug abuse within the past 1 year;
* Has a history of confirmed neurological or mental disorders, such as epilepsy, dementia; or poor compliance;
* Is pregnant or breastfeeding;
* Other reasons disqualifying the entering of this study based on the evaluation of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 24 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
Disease Control Rate (DCR) | 24 months
Duration of Response (DOR) | 24 months
Progress Free Survival (PFS) | 24 months
Overall Survival (OS) | 36 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hunan Cancer Hospital, Changsha
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan